CLINICAL TRIAL: NCT03395821
Title: Comparison Between Exclusive Surgical Training Versus Virtual Reality Plus Traditional Training in Surgical Skills of Residents of Obstetrics and Gynecology
Brief Title: Traditional Versus Virtual Reality for Surgical Skills for ObGyn Residents
Acronym: SIMUTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Ricardo Francalacci Savaris, Professor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-0365
Record Dates: First submitted 2017-12-27; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Gynecologic Disease
Keywords: competency-based education; gynecology; laparoscopy; resident education; simulation; surgical curriculum
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: Two groups will be compared according to their surgical skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional training (Active Comparator): Residents will receive the traditional training for laparoscopic surgery according to their residency program.
  Interventions: Behavioral: Conventional training
- Virtual Reality+conventional training (Experimental): Residents will receive 12 weeks of virtual training for laparoscopy and their traditional training for laparoscopic surgery according to their residency program.
  Interventions: Behavioral: Virtual Reality+conventional training

INTERVENTIONS:
Behavioral: Conventional training — traditional training according to residency program
  Arms: Conventional training
Behavioral: Virtual Reality+conventional training — virtual reality training+traditional training using virtual reality
  Arms: Virtual Reality+conventional training

SUMMARY:
This study will verify if a comprehensive laparoscopic curriculum using virtual reality demonstrates skills transfer to the operating room, compared to the traditional teaching method.

DETAILED DESCRIPTION:
Second-year residents from different programs of residency in obstetrics and gynecology in Porto Alegre, RS, Brazil, will be invited to participate in this study. they will be randomized to receive a comprehensive training in laparoscopy using modern virtual reality program or the traditional method of training according to their residency program. After 12 weeks of training, they will finish their training and they will perform advanced laparoscopic surgery in the simulator according to their specific needs, for example, salpingectomy, oophorectomy advanced laparoscopic suture or hysterectomy. Data generated from the simulator program will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* residents in obstetrics and gynecology that are about to finish their second-year program

Exclusion Criteria:

* refuse to participate

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficiency of technical skills (%) | 12 weeks
  The software analyzes the percentage of time the needle-holders' ends are kept outside the operative field (%); total number of entrance and exit points through which the needle has passed; total aggressive tissue handling; total amount of strain applied to tissue during needle passages; total needle loading time; total number of completed knots; total number of needle loadings; total number of needle passages; total number of stitches; total time the needle-holders' ends are kept outside the predefined operative field; total time to accomplish the suture; Total time to form a knot. For salpingectomy: efficiency of cautery (%); number of non-cauterized bleeding; number of serious complications: possible damage to vital structures; safe cautery (%); the time cautery is applied without appropriate contact with adhesions; total number of applied clips.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro T Cavazzola, MD,PhD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shirai Y, Yoshida T, Shiraishi R, Okamoto T, Nakamura H, Harada T, Nishikawa J, Sakaida I. Prospective randomized study on the use of a computer-based endoscopic simulator for training in esophagogastroduodenoscopy. J Gastroenterol Hepatol. 2008 Jul;23(7 Pt 1):1046-50. doi: 10.1111/j.1440-1746.2008.05457.x. Epub 2008 Jun 28. PMID 18554236
- [Result] Palter VN, Grantcharov TP. Individualized deliberate practice on a virtual reality simulator improves technical performance of surgical novices in the operating room: a randomized controlled trial. Ann Surg. 2014 Mar;259(3):443-8. doi: 10.1097/SLA.0000000000000254. PMID 24503910
- [Result] Shore EM, Grantcharov TP, Husslein H, Shirreff L, Dedy NJ, McDermott CD, Lefebvre GG. Validating a standardized laparoscopy curriculum for gynecology residents: a randomized controlled trial. Am J Obstet Gynecol. 2016 Aug;215(2):204.e1-204.e11. doi: 10.1016/j.ajog.2016.04.037. Epub 2016 Apr 27. PMID 27131588